CLINICAL TRIAL: NCT02972099
Title: The Psychological Effects of Transcutaneous Pulsed Radiofrequency (TcPRF) in Patients With Emotional Stress
Brief Title: Pulsed Radiofrequency for Emotional Stress
Acronym: TcPRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2015-12
Record Dates: First submitted 2016-11-18; First posted 2016-11-23 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TcPRF Group (Experimental): According to the standard application of the device, for the PRF procedure one 5 x 13 cm skin electrode will be placed over the forehead, the other one over the posterior aspect of the neck. PRF with a duty load of 14.8 msec/sec and an average pulse frequency of 5.11 Hz will be applied for 25min. The voltage will be set to generate a current of 1 A.
  Voltage and impedance will be monitored continuously during treatment and if necessary the voltage will be corrected to ensure the proper current.
  Interventions: Device: TcPRF
- Placebo Group (Placebo Comparator): The setup will be made as for active treatment but no current will be delivered. The patients will not be able to feel any difference to the real treatment.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: TcPRF — Transcutaneous Pulsed Radiofrequency is a method that is widely used for control of pain. There are no known complications. In this study a Radiofrequency generator will be used that has a separate outlet for transcutaneous use. It is used in the daily clinical practice in the Pain Center of the Swiss Paraplegic Center.
  Other Names: TOP Lesion Generator TLG-10 (TOP Corporation - Tokyo, Japan)
  Arms: TcPRF Group
Device: Placebo — In the Placebo Treatment, no current will be delivered. Since no sensations are produced by TcPRF treatment the patients won't recognize the difference.
  Other Names: TOP Lesion Generator TLG-10 (TOP Corporation - Tokyo, Japan)
  Arms: Placebo Group

SUMMARY:
The objective of the study is to assess the short-term and long-term effects of transcutaneous pulsed radio frequency treatment on the physiological status, subjective well-being, and on the intensity of pain. Category A Transcutaneous Pulsed Radiofrequency is a method that is widely used for control of pain. There are no known complications. In this study a Radiofrequency generator will be used that has a separate outlet for transcutaneous use. Patients will be recruited within the clinic population of patients.

DETAILED DESCRIPTION:
Data will be assessed in at three times, the baseline testing, the first and the second follow-up meeting (+2-4 days of intervention; as well as + 40 days via post/email)

The inclusion criteria are: Inclusion:

* age 18 - 65
* chronic pain (Duration of three Months or more) patients of the Pain Center Nottwil, Swiss Paraplegic Center

The following criteria will lead to an exclusion of the study:

* severe medical issues, such as cancer or comparable diseases
* severe mental disorders such as severe depression or schizophrenia
* patients with pacemakers or with atrial fibrillation
* Women who are pregnant or breast-feeding The primary outcome assessed is the physiological status, assessed by the heart rate variability (HRV). Secondary outcomes are the subjective well-being, as assessed by the "Marburger questionnaire regarding habitual well-being" (FW-7) questionnaire as well as the intensity of pain, as assessed by the numeric rating scale for pain intensity (NRS) score and by a 7-point Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 65
* chronic pain (Duration of three Months or more) patients of the Pain Center, Swiss Paraplegic Center, Nottwil

Exclusion Criteria:

* severe medical issues, such as cancer or comparable diseases
* severe mental disorders such as severe depression or schizophrenia
* patients with pacemakers or with atrial fibrillation
* Women who are pregnant or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Physiological status - Change between Baseline and Follow-up 1 | Baseline; Follow-up 1 (+2-4 days)
  physiological status, assessed by the heart rate variability (HRV)

SECONDARY OUTCOMES:
Subjective Wellbeing - Change between Baseline and Follow-up 1 & 2 | Baseline; Follow-up 1 (+2-4 days); Follow-up 2 (+40 days by post)
  Secondary outcome is the subjective well-being, as assessed by the FW-7 questionnaire
Intensity of pain - Change between Baseline and Follow-up 1 & 2 | Baseline; Follow-up 1 (+2-4 days); Follow-up 2 (+40 days by post)
  the intensity of pain is assessed by the Numeric Rating Scale for pain (NRS) score by a 7-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lacher, Dr. phil., Principal Investigator — Pain Center, Swiss Paraplegic Center
Locations (1):
- Pain Center, Swiss Paraplegic Center, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No